CLINICAL TRIAL: NCT02126878
Title: Prospective, Randomized, Double-blinded Comparison of Steroid Dosages on the Efficacy of Trochanteric Bursa Injection
Brief Title: Comparison of Steroid Dosages on the Efficacy of Trochanteric Bursa Injection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: West Virginia University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1401174207
Record Dates: First submitted 2014-04-26; First posted 2014-04-30 (Estimated); Results first posted 2021-01-20 (Actual); Last update posted 2021-10-19 (Actual); Status verified 2021-09

CONDITIONS: Bursitis
MeSH Terms: conditions — Bursitis | interventions — Triamcinolone Acetonide

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Kenalog 20mg (Active Comparator): 20mg/ 2ml and local anesthetic
  Interventions: Drug: Kenalog
- Kenalog 40mg (Active Comparator): 40mg/ 2ml with local anesthetic
  Interventions: Drug: Kenalog
- Kenalog 80mg (Active Comparator): 80mg/ 2ml and local anesthetic
  Interventions: Drug: Kenalog

INTERVENTIONS:
Drug: Kenalog

SUMMARY:
Inflammation of the trochanteric bursa is a common cause of hip pain. A bursa is a closed fluid filled sac or sac-like cavity found between tissues that function as a gliding surface to reduce friction. Bursitis is the inflammation of the bursa. Inflammation between the trochanteric process of the femur and gluteus medius tendon/ iliotibial tract is the cause of trochanteric bursitis. Several treatments exist for trochanteric bursitis, including a local steroid injection. The injection consists of a mixture of local anesthetic and steroid medications. The steroid is routinely mixed with a local anesthetic. The anesthetic acts to diluent the steroid as well as act as a pain reliever. Various steroid preparations have been used, at varying doses, for trochanteric bursitis. The steroid preparation, triamcinolone is commonly used for various reasons. Besides the procedure associated and injection site risks, risks associated with the use of steroids, though rare, exist. Short term, the steroid can raise blood sugar levels and should be used with caution and be appropriately monitored in diabetics. Additionally, the steroid can suppress the immune system. Long-term risks are related to the dose and frequency of use. These risks include thinning of the skin, easy bruising, weight gain, elevated blood pressure, cataract formation, thinning of bones and joints. Studies have shown the effectiveness of local steroid injections for trochanteric bursitis. Unfortunately, there is limited data on the ideal dose of the steroid preparation. Triamcinolone of 40mg/ mL is commonly used, but, studies have shown effectiveness at various doses, ranging 20 to 160 mg/mL. The aim of this study is to evaluate and compare the effectiveness of local steroid injections of various steroid dosages for the treatment of trochanteric bursitis.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of trochanteric bursitis
2. 18 years of age or older when written informed consent is obtained
3. Signed institutional review board approved informed consent form

Exclusion Criteria:

1. Meets any contraindication for treatment
2. Allergy to triamcinolone, lidocaine
3. Previous surgery to bursa
4. Coagulopathy
5. Active Infection
6. Currently diagnosed with cognitive impairment, or exhibits any characteristic, that would limit study candidate's ability to assess pain relief or complete study assessments

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2014-04; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- West Virginia University Hospitals, Morgantown, West Virginia, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was ended and the PI has left the institution. The numbers presented are what was initially entered by the research team. From data available, 120 participants were enrolled on the study; no information about those participants could be located. No other data could be located and it cannot be determined which arm the120 participants were enrolled in or if they completed the study.
Groups:
- Kenaglog 20mg: 20mg/ 2ml and local anesthetic
  Kenalog
- Kenalog 40mg: 40mg/ 2ml with local anesthetic
  Kenalog
- Kenalog 80mg: 80mg/ 2ml and local anesthetic
  Kenalog
Period: Overall Study
Arm/Group | Kenaglog 20mg | Kenalog 40mg | Kenalog 80mg
Started | 0 | 0 | 0
Completed | 0 | 0 | 0
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The study was ended and the PI has left the institution. No results information is available, all efforts were to made to retrieve results information, but were unsuccessful. No study data is available.
Groups:
- Total: Total of all reporting groups
Arm/Group | Kenaglog 20mg | Kenalog 40mg | Kenalog 80mg | Total
Number analyzed (Participants) | 0 | 0 | 0 | 0
Age, Categorical
Sex: Female, Male
Race and Ethnicity Not Collected — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Pain Intensity Measured on Visual Analog Scale and Percent Improvement
Time Frame: 3 month
Population: as for baseline characteristics
Arm/Group | Kenaglog 20mg | Kenalog 40mg | Kenalog 80mg
Number analyzed (Participants) | 0 | 0 | 0

2. Secondary Outcome: Disability Measured on Becks Disability Scale
Time Frame: Baseline, 1 month, 3 month
Population: as for baseline characteristics
Arm/Group | Kenaglog 20mg | Kenalog 40mg | Kenalog 80mg
Number analyzed (Participants) | 0 | 0 | 0

3. Secondary Outcome: Safety, Adverse Affects
Time Frame: 1 month,3 months
Population: as for baseline characteristics
Arm/Group | Kenaglog 20mg | Kenalog 40mg | Kenalog 80mg
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Description: The study was ended and the PI has left the institution. No results information is available, all efforts were to made to retrieve results information, but were unsuccessful. No study data is available.
Arm/Group | Kenaglog 20mg | Kenalog 40mg | Kenalog 80mg
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
This study is considered to be completed, because before leaving the institution the PI indicated the study status as completed and entered that actual enrollment number of 120 participants. No other information could be located or obtained for the study and therefore no specific results information can be included. The study status as completed and actual enrollment number of 120 participants should be considered an accurate representation of all available study information.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes